CLINICAL TRIAL: NCT05161741
Title: Research on Human Insulin rDNA (Insuget) Safety and Efficacy in Patients With Type 2 Diabetes Mellitus
Brief Title: Research on Human Insulin rDNA Safety and Efficacy in Patients With Type 2 Diabetes Mellitus
Acronym: RISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Getz Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTZ-DM-004-21
Record Dates: First submitted 2021-12-16; First posted 2021-12-17 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2021-12

CONDITIONS: Adverse Drug Event; Effect of Drug; Type 2 Diabetes Treated With Insulin
Keywords: Insulin; Type 2 Diabetes mellitus; Safety; Efficacy
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Uncontrolled diabetes requiring Insulin (Experimental)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Human rDNA Insulin (Insuget, local brand of Getz Pharma)

SUMMARY:
Objective: To evaluate the safety and efficacy of Human Insulin rDNA (Insuget) in patients with Type II Diabetes Mellitus.

Study Design: Open-label, prospective, observational, single arm, multi-center, post-marketing surveillance study.

Sample size: The estimated target sample size is n=230. Study duration: 12 months (data lock point will be completion of 6 months' follow-up from the time of last patient's enrollment date)

After recruitment, patient is supposed to have three visits for follow-ups. Visit 1: 4 to 6 weeks of initiation of therapy. Visit 02: At 12 weeks of initiation of therapy. Visit 03: At 24 weeks of initiation of therapy.

* Primary (SAFETY Outcomes):

  * Frequency of adverse events during the course of study follow-up.
  * Frequency of serious adverse events.
* SECONDARY OUTCOME MEASURES (EFFICACY ENDPOINTS)

  * Change from baseline in HbA1c% to the last-observation.
  * Change from baseline in fasting plasma glucose to the last- observation on treatment

Ethical consideration:

The ethical approval of study is taken from an independent ethics committee. The study will be conducted in compliance with the protocol, good clinical practices (GCP), the ethical principles that have their origin in the Declaration of Helsinki and the applicable regulatory requirements.

DETAILED DESCRIPTION:
OBJECTIVE To evaluate the safety and efficacy of Human Insulin rDNA (Insuget) in patients with Type II Diabetes Mellitus.

METHODOLOGY:

STUDY DESIGN:

Open-label, prospective, observational, single arm, multi-center, post-marketing surveillance study.

SAMPLE SIZE As per cited literature, the reported hypoglycemia rate was 41% in patients who underwent treatment of Human Regular Insulin.

Considering 10% increase of hypoglycemia incidence in current study from the reference literature and keeping 95% confidence level, 5% margin of error and 80% power of study, the calculated sample size is n=191. After adding 20% attrition rate, the target enrollment would be n=230.

NUMBER OF SITES Total 04-05 sites.

STUDY DURATION 10-12 months (data lock point will be completion of 6 months' follow-up from the time of last patient's enrollment date)

SAMPLING TECHNIQUE A non-probability consecutive sampling method will be used to screen patients as per study eligibility criteria.

LABORATORY TESTING:

Reputable laboratory is considered for testing of diabetes patients i.e. HbA1c and FBG. The certified clinical lab will be responsible for receiving and analyzing clinical sample.

HbA1c and FBG readings would be recorded within ±10 days of the follow up visit and FBG ±03 day of the follow up visit or average of last three reading in the diary reported by patient, respectively.

SCREENING / BASELINE VISIT After taking the informed consent, the patient will be screened as per the defined criteria and further will be initiated on Insuget (Human Insulin rDNA).

The following data will be recorded on the baseline visit.

* Date of visit
* Inclusion & Exclusion criteria will be evaluated for enrollment
* Demographic data: Age (years), Gender
* Physical parameters i-e weight (kg), height (inches), BMI (Kg/m2)
* Duration of Diabetes (years)
* Smoking status: Yes / No
* Education Level: Graduate or above / Secondary or below / No Formal Education
* Blood pressure readings (mm/Hg)
* Concomitant Disease and Therapy Details

Laboratory Investigations:

* HbA1c and FBS

  • Insulin use status
* Insulin naïve or already on insulin therapy with dose/frequency details

VISIT 1 (1st follow-up visit; after 4 to 6 weeks of initiation of therapy)

Each patient will have a unique study patient number; the following information will be recorded at the 1st follow-up visit:

* Date of visit
* Physical parameters i-e weight (kg)
* Blood pressure

Laboratory Investigations:

o FBS

Safety Evaluation i-e Hypoglycemia; Symptoms of Hypoglycemia: Headache, Feeling of Hunger, Drowsiness, Blurred Vision, Sweating, Nausea, Confusion, Dizziness, Tachycardia, Tremor and others.

* Hypokalemia; Muscle Cramps, Weakness, Irregular Heart Beat and others
* Injection Site Related Adverse Events; Pain, Redness, Irritation, Lipodystrophy and others.

Review of Patient Diary and reporting Self-monitoring blood glucose: Last three readings average will be taken for fasting blood glucose.

Reports of any serious adverse events leading to hospitalization i-e severe hypoglycemia.

VISIT 2 (2nd follow-up visit; after 3 months of initiation of therapy)

Each patient will have a unique study patient number; the following information will be recorded at the 1st follow-up visit:

* Date of visit
* Physical parameters i-e weight (kg)
* Blood pressure

Laboratory Investigations:

-HbA1c and FBS

Safety Evaluation i-e

* Hypoglycemia; Symptoms of Hypoglycemia: Headache, Feeling of Hunger, Drowsiness, Blurred Vision, Sweating, Nausea, Confusion, Dizziness, Tachycardia, Tremor and others.
* Hypokalemia; Muscle Cramps, Weakness, Irregular Heart Beat and others.
* Injection Site Related Adverse Events; Pain, Redness, Irritation, Lipodystrophy and others.

Review of Patient Diary and reporting Self-monitoring blood glucose: Last three readings average will be taken for fasting blood glucose.

Reports of any serious adverse events leading to hospitalization i-e severe hypoglycemia.

VISIT 3 (3rd follow-up visit at 6 months of initiation of therapy)

Each patient will have a unique study patient number; the following information will be recorded at the 1st follow-up visit:

* Date of visit
* Physical parameters i-e weight (kg)
* Blood pressure

Laboratory Investigations:

-HbA1c and FBS

Safety Evaluation i-e

* Hypoglycemia; Symptoms of Hypoglycemia: Headache, Feeling of Hunger, Drowsiness, Blurred Vision, Sweating, Nausea, Confusion, Dizziness, Tachycardia, Tremor and others.
* Hypokalemia; Muscle Cramps, Weakness, Irregular Heart Beat and others.
* Injection Site Related Adverse Events; Pain, Redness, Irritation, Lipodystrophy and others.

Review of Patient Diary and reporting

* Self-monitoring blood glucose: Last three readings average will be taken for fasting blood glucose.
* Reports of any serious adverse events leading to hospitalization i-e severe hypoglycemia.

STUDY TREATMENT After obtaining consent and baseline assessment, the patient will be advised to start Insuget (Human Insulin rDNA) and will be assessed in follow-up visits as per the defined parameters.

DOSE & FREQUENCY OF STUDY TREATMENT The investigator will recommend the dose of Insuget 70/30 (Local Insulin brand) and/or Insuget N (Local Insulin brand) and/or Insuget R (Local Insulin brand) as per standard clinical practices to meet the daily requirements of study patients.

The drug frequency will be at the discretion of the treating physician. Patients included in the study will be administered treatment according to the standard guidelines.

CONCOMITANT TREATMENT Concomitant treatment for hypertension, dyslipidemia, and other associated diseases will be continued as per the physician's discretion and/or according to the standard guidelines. Similarly, other treatments can be initiated during the course of the study as and when needed. All concomitant medications must be documented.

DATA COLLECTION An electronic data capture system will be used for this study. An electronic database will be designed to record the data required by the protocol and collected by the investigator. All personal data will be coded with a unique number; the researcher will securely keep codes at the research site. Potential participant will have to sign the consent to take part in the study but all personal data collected during the study will be dealt with strict confidentiality and will be used for the research in coded form.

Coded data will be transferred and processed following applicable laws, regulations protecting processing, and transfer of coded data. As per data protection laws and regulations, patients may be titled to access, rectify and ask for the deletion of their personal data via their doctors who are the only person to know the correspondence between the participant number and identity. Personal data will be kept until the publication of the results of the study and will then be archived.

DISCONTINUATION OF TREATMENT Any significant adverse event, which leads to discontinuation from the study treatment. The time and reason for discontinuation will be recorded in the CRF.

DATA MANAGEMENT AND STATISTICAL ANALYSIS Statistical analyses will be performed using SPSS version-22. Mean ±standard deviation will be calculated for continuous variables like age, height, weight, BMI, blood pressure, duration of diabetes, HbA1c and FBS whereas categorical variables will be presented as frequencies and percentages (gender, smoking status, education level, comorbidities, adverse events, etc). Age will be stratified to evaluate the association of reported adverse events with age group and other categorical variable will be assessed through chi-square test. ANOVA will be applied to determine the reduction of HbA1c, FBS, Weight, BMI and Blood Pressure from baseline to 6 months follow-up. A normality test will be done for consideration of parametric or non-parametric application of significance tests. P-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written informed consent.
* Type 2 diabetic males & females with age 18 & above years.
* HbA1c: 7.0% and above.
* Patients with uncontrolled Diabetes after intervention of lifestyle modifications plus oral and/or insulin therapy.

Exclusion Criteria:

* Known type 1 diabetes mellitus patients.
* History of severe hypoglycemia (<70mg/dL)
* History of hypersensitivity to any of the active or inactive ingredients of the insulin preparations used in the trial, and/or history of significant allergic drug reactions.
* Presence of severe diabetes complications.
* History of renal and/or hepatic dysfunctions.
* Patients who have been admitted to the hospital in the past 3 months for diabetic ketoacidosis (DKA) and hyperosmolar hyperglycemic state.
* History of acute coronary syndrome or stroke.
* Pregnant or lactating females.
* History of Acute psychiatric disorder or exacerbation of chronic psychiatric disorder.
* History or presence of a medical condition or disease that in the investigator's opinion would embarrass glycemic control and completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events, serious adverse events during the course of study follow-up | 6 months
  Drug safety
Change from baseline in HbA1c% to the last-observation | 6 months
  Drug efficacy
Change from baseline in fasting plasma glucose to the last- observation on treatment | 6 months
  Drug efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Social Security Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2008 Jan;31 Suppl 1:S55-60. doi: 10.2337/dc08-S055. No abstract available. PMID 18165338
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Turner RC, Cull CA, Frighi V, Holman RR. Glycemic control with diet, sulfonylurea, metformin, or insulin in patients with type 2 diabetes mellitus: progressive requirement for multiple therapies (UKPDS 49). UK Prospective Diabetes Study (UKPDS) Group. JAMA. 1999 Jun 2;281(21):2005-12. doi: 10.1001/jama.281.21.2005. PMID 10359389
- [Background] Wright A, Burden AC, Paisey RB, Cull CA, Holman RR; U.K. Prospective Diabetes Study Group. Sulfonylurea inadequacy: efficacy of addition of insulin over 6 years in patients with type 2 diabetes in the U.K. Prospective Diabetes Study (UKPDS 57). Diabetes Care. 2002 Feb;25(2):330-6. doi: 10.2337/diacare.25.2.330. PMID 11815505